CLINICAL TRIAL: NCT03918434
Title: Efficacy of a Locoregional Anesthesia Technique During High Energy Extracorporeal Shock Wave Therapy for Painful Foot Disease: a Pilot Study
Brief Title: Efficacy of a Locoregional Anesthesia Technique During Shock Wave Therapy
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, SPINAZZOLA GIORGIA, Medical doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 200319/1
Record Dates: First submitted 2019-04-06; First posted 2019-04-17 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Achilles Tendinopathy; Plantar Fascitis
Keywords: tibial nerve block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Plantar fasciitis and the chronic Achilles tendinopathy are the most common causes of heel pain. The term "plantar fasciitis" implies an inflammatory condition by the suffix "itis". However, various lines of evidence indicate that this disorder is better classified as "fasciosis" or "fasciopathy", as heel pain associated with degenerative changes in the fascia and atrophy of the abductor minimi muscle. High energy shock wave therapy (HESWT) has been proposed as a potential method of treating patients with chronic disease without the need to stop weightbearing. Often a crucial complication of HESWT is the appearance of pain with the subsequent interruption of the procedure. The consequences are a reduced patient compliance, need of a deep sedation and more sessions for the treatment.

Frequently, topic anesthesia (TA) (as EMLA) is applied during the therapy to decrease the pain HESWT-induced and enable sham treatment. Multiple publications focused on the evaluation of a clinically relevant eﬀect of shock wave application on plantar heel pain, either of HESWT, applied in a single session with local or regional anesthesia or of low energy HESWT, applied repetitively without local anesthesia.

Rompe JD and colleagues have demonstrated that the therapeutic success rate of HESWT with TA is significantly smaller than without TA even after 3 months. Probably, the use of anesthetic topically applied can reduce the efficacy of HESWT for increased impedance. To date, many patients interrupted the HESWT for moderate-severe pain. Consequently, this therapy, which generally is administered in three sessions, required a prolongation of procedure up to six sessions.The clinical application of Posterior Tibial nerve block (already widely used in operating room) during HESWT applied in Orthopedic Day Hospital could offer the possibility to minimize the patient discomfort and to give the therapeutic doses just in few HESWT sessions, reducing the hospital access of outpatients for the treatments and the costs related to prolonged treatment caused by pain. Furthermore, this anesthetic approach could make patients tolerate majorated doses of HESWT in few sessions, with high effectiveness of procedure after several months.

DETAILED DESCRIPTION:
The aim of this pilot prospective observational study is to allow outpatients with chronic Achilles tendinopathy and plantar fasciitis to reduce the pain during HEWST. The study will be focused on the evaluation of a posterior tibial nerve block efficacy in patients who discontinued the first application of HESWT due to surge of moderate-severe pain.

Objectives of the study Primary objective The primary objective of the study is to observe a 40% reduction in Numerical Rating Scale (NRS) from baseline (T0) to T1 during HESWT.

Secondary objectives: evaluation of the number of patients that are able to complete a single session with Posterior tibial nerve block (usually, without Posterior tibial nerve block, 40% of patients can not complete the session); evaluation of the number of sessions required to complete successfully the treatment (usually, without Posterior tibial nerve block, the number of sessions required to complete successfully the treatment is 6); evaluation of the efficacy of HESWT (American Orthopedic Foot and Ankle Society Score - AOFAS, performed 1 month from the end of treatment).

Design of the study This is an observational, pilot, prospective, cohort study. It will be conducted in Orthopedic Day Hospital Ward of "Fondazione-Policlinico Universitario A. Gemelli IRCCS" of Rome. The planned duration of the study is 6th months and the proposed sample size is N:21.

Materials and Methods The enrollment starts after the patient interrupt his/her first HESWT treatment (T0) because the pain is unbearable with NRS>5. Before the second HESWT session (T1) patients will receive the posterior tibial nerve block (PTNB) under ultrasound control. This anesthetic procedure will be repeated for every subsequent HESWT session. After each treatment, the patient will be monitored in Orthopedic Day hospital ward for about 2 hours or until complete sensitive recovery. At the end of each session the patient will be asked to express his/her pain intensity using the NRS.

The anesthetic procedure With the patient lying supine and the foot externally rotated, an expert anesthesiologist will perform the PTNB with echo guided, finding the posterior tibial nerve between the middle and the distal third of the leg, about 6-8 cm proximally to the tibial malleolus. Once the nerve will be identified, the needle (70 millimeters long, 22 gouge, UPC Polymedic) will insert in-plain and after careful aspiration mepivacaine 1 % (3-4 ml) will injected.

Measurements Intensity of pain at the end of each procedure will be measured by Numerical Rating Scale (NRS) between 0 and 10 points, where Zero usually represents 'no pain at all' whereas ten represents 'the worst pain ever possible.

Evaluation of patient's adherence to the treatment, will be detected as the number of patients that manage to complete the session The sensitive block duration will be evaluated by pinprik test (defined as a test for cutaneous pain receptors. A small, clean, sharp object such as a pin or needle is gently applied to the skin and the patient is asked to describe the sensation. One must be certain the patient is reporting the sensation of pain rather than that of pressure.) The efficacy of HESWT will be evaluated by American Orthopedic Foot and Ankle Society Score (AOFAS) after 1 month from the end of treatment. Each measure of AOFAS is comprised of nine questions and cover three categories: Pain (40 points), function (50 points) and alignment (10 points). These are all scored together for a total of 100 points.

Inclusion criteria

Patients will be enrolled if they present all of the following criteria:

History of Chronic Achilles tendinopathy and/or plantar fasciitis at least 6 months long Unsatisfying subjective result (Numeric Rating Scale (NRS) score persistently ≥ 4 points for pain during the ﬁrst few steps of walking in the morning) after at least 6 months after ≥ 3 of the following 5 conventional therapy programs: ≥ 4 weeks of physical therapy; ≥4 weeks course of non-steroidal anti-inﬂammatory medications HEWST indication Application of HESWT at 1500 shock waves with energy of 16 Ky First treatment discontinued for surge of pain (numeric rating scale > 5) Exclusion criteria Patient < 18 years Peripheral circulatory disorders Arthrosis of the foot or ankle, as conﬁrmed by X-ray diagnosis Skin lesions of the foot Allergy to local anesthetic Neurologic abnormality (changes of deep tendon reﬂexes, motor or sensory deﬁcit) Routinely consumption of analgesics or history of analgesic consumption within 24 hours prior to therapy.

Statistical Plan Sample size determination As a pilot study, no data is available in the literature. The proposed sample size is N:21 patients. This dimension provides a power of 0.99, with confidence level = 0.05 of detecting a 40% reduction in the NSR score from T0 to T1.

Statistical analysis The sample will be described in its clinical and demographic features using descriptive statistics techniques. Quantitative variables will be described using the following measures: minimum, maximum, range, mean and standard deviation. Qualitative variables will be summarized with absolute and percentage frequency tables. Normality of data will be verified using the Kolmogorov-Smirnov test.

The primary objective will be achieved performing a Student's T test for paired sample.

The proportion of patients that are able to complete a single session with Posterior tibial nerve block will be evaluated and compared to the same proportion in patients without Posterior tibial nerve block (40% of patients can not complete the session); The mean and median number of sessions required to complete successfully the treatment will be calculated.

The evaluation of HESWT efficacy will be performed via the AOFAS score, comparing proportions using the Chi squared test.

Possible comparisons will be performed with the Student T test for paired sample (if data are normally distributed) or with the Wilcoxon test (for non normal distribution). Comparison of categorical data will be performed using a Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* • History of Chronic Achilles tendinopathy and/or plantar fasciitis at least 6 months long

  * Unsatisfying subjective result (Numeric Rating Scale (NRS) score persistently ≥ 4 points for pain during the ﬁrst few steps of walking in the morning) after at least 6 months after ≥ 3 of the following 5 conventional therapy programs: ≥ 4 weeks of physical therapy; ≥4 weeks course of non-steroidal anti-inﬂammatory medications
  * HESWT indication
  * Application of HESWT at 1500 shock waves with energy of 16 Ky
  * First treatment discontinued for surge of pain (numeric rating scale [NRS] > 5)

Exclusion Criteria:

* • Patient < 18 years

  * Peripheral circulatory disorders
  * Arthrosis of the foot or ankle, as conﬁrmed by X-ray diagnosis
  * Skin lesions of the foot
  * Allergy to local anesthetic
  * Neurologic abnormality (changes of deep tendon reﬂexes, motor or sensory deﬁcit)
  * Routinely consumption of analgesics or history of analgesic consumption within 24 hours prior to therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, with History of Chronic Achilles tendinopathy and/or plantar fasciitis at least 6 months long, who interrupt his/her first HESWT treatment (T0) because the pain is unbearable with NRS>5.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Number of patients who reported a reduction of pain during High Energy Shock Wave Therapy with posterior nerve block | 6th months
  The primary objective of the study is to observe a 40% reduction in Numerical Rating Scale before and after posterior tibial nerve block during shock wave therapy. Intensity of pain at the end of each procedure will be measured by Numerical Rating Scale (NRS) between 0 and 10 points, where Zero usually represents 'no pain at all' whereas ten represents 'the worst pain ever possible.

SECONDARY OUTCOMES:
Number of patients who completed the session of shock wave therapy | 6th months
  evaluation of the number of patients that are able to complete a single session with Posterior tibial nerve block
Number of shock wave sessions | 6th months
  evaluation of the number of sessions required to complete successfully the treatment
Number of patients with clinical efficacy of shock wave therapy evaluated by American Orthopedic Foot and Ankle Society Score (AOFAS) | 7th months
  evaluation of the efficacy of High Energy Shock Wave Therapy after 1 month from the end of treatment by American Orthopedic Foot and Ankle Society Score (AOFAS). Each measure of AOFAS is comprised of nine questions and cover three categories: Pain (40 points), function (50 points) and alignment (10 points). These are all scored together for a total of 100 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Spinazzola Giorgia, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furia JP. High-energy extracorporeal shock wave therapy as a treatment for insertional Achilles tendinopathy. Am J Sports Med. 2006 May;34(5):733-40. doi: 10.1177/0363546505281810. PMID 16627628
- [Background] Schmitz C, Csaszar NB, Rompe JD, Chaves H, Furia JP. Treatment of chronic plantar fasciopathy with extracorporeal shock waves (review). J Orthop Surg Res. 2013 Sep 3;8:31. doi: 10.1186/1749-799X-8-31. PMID 24004715
- [Background] Notarnicola A, Maccagnano G, Tafuri S, Fiore A, Margiotta C, Pesce V, Moretti B. Prognostic factors of extracorporeal shock wave therapy for tendinopathies. Musculoskelet Surg. 2016 Apr;100(1):53-61. doi: 10.1007/s12306-015-0375-y. Epub 2015 May 16. PMID 25982090
- [Background] Speed CA, Nichols D, Wies J, Humphreys H, Richards C, Burnet S, Hazleman BL. Extracorporeal shock wave therapy for plantar fasciitis. A double blind randomised controlled trial. J Orthop Res. 2003 Sep;21(5):937-40. doi: 10.1016/S0736-0266(03)00048-2. PMID 12919884
- [Background] Aqil A, Siddiqui MR, Solan M, Redfern DJ, Gulati V, Cobb JP. Extracorporeal shock wave therapy is effective in treating chronic plantar fasciitis: a meta-analysis of RCTs. Clin Orthop Relat Res. 2013 Nov;471(11):3645-52. doi: 10.1007/s11999-013-3132-2. Epub 2013 Jun 28. PMID 23813184
- [Background] Lou J, Wang S, Liu S, Xing G. Effectiveness of Extracorporeal Shock Wave Therapy Without Local Anesthesia in Patients With Recalcitrant Plantar Fasciitis: A Meta-Analysis of Randomized Controlled Trials. Am J Phys Med Rehabil. 2017 Aug;96(8):529-534. doi: 10.1097/PHM.0000000000000666. PMID 27977431
- [Background] Rompe JD, Meurer A, Nafe B, Hofmann A, Gerdesmeyer L. Repetitive low-energy shock wave application without local anesthesia is more efficient than repetitive low-energy shock wave application with local anesthesia in the treatment of chronic plantar fasciitis. J Orthop Res. 2005 Jul;23(4):931-41. doi: 10.1016/j.orthres.2004.09.003. PMID 16023010
- [Background] Klonschinski T, Ament SJ, Schlereth T, Rompe JD, Birklein F. Application of local anesthesia inhibits effects of low-energy extracorporeal shock wave treatment (ESWT) on nociceptors. Pain Med. 2011 Oct;12(10):1532-7. doi: 10.1111/j.1526-4637.2011.01229.x. Epub 2011 Sep 14. PMID 21917114
- [Result] Rompe JD. Plantar fasciopathy. Sports Med Arthrosc Rev. 2009 Jun;17(2):100-4. doi: 10.1097/JSA.0b013e3181a3d60e. PMID 19440137